CLINICAL TRIAL: NCT02549872
Title: Dementia Phenotypes in Primary Care, Hospital, and National Mortality Registries: a Cohort Study in Linked Electronic Health Records
Brief Title: Dementia Phenotypes in Primary Care, Hospital, and National Mortality Registries
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: University of Edinburgh (Other); University of Leeds (Other); Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Harry Hemingway, Professor of Epidemiology and Public Health, University College, London
Other Study IDs: 15_138
Record Dates: First submitted 2015-09-03; First posted 2015-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Dementia
Keywords: Dementia; Validity; Mortality; Electronic health records
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Dementia: Patients with a recorded diagnosis of dementia in primary or secondary care
  Interventions: Other: This is not an intervention study
- Non-dementia: Patients without a recorded diagnosis of dementia in primary or secondary care
  Interventions: Other: This is not an intervention study

INTERVENTIONS:
Other: This is not an intervention study — This study is based on the retrospective analysis of linked electronic health records.

SUMMARY:
Most patients with dementia in the UK use their local hospitals and general (family) practices throughout their illness. Linked electronic health records from primary care, hospital and death certificates records therefore provide useful information about the diagnosis and prognosis of patients who develop dementia.

In this study we will assess the validity of dementia diagnoses in linked primary care, hospital and death records, by examining the timing of important health transitions in patients with recorded dementia, and we will estimate the lifetime risk of recorded dementia in different age and sex groups

DETAILED DESCRIPTION:
Dementia is a clinical syndrome with insidious onset that is difficult to diagnose in its earliest stages. Presentation to healthcare depends not only upon the rates of disease progression, but also on social support, recognition by clinicians, and patients' and carers' fear of diagnosis. Maintaining complete follow up in cohorts of patient with dementia is difficult, because patients with dementia are frequently lost to follow up.

Most patients with dementia in the UK use their local hospitals and general (family) practices throughout their illness. Linked electronic health records from primary care, hospital and death certificates records should therefore provide useful information about the diagnosis and prognosis of patients who develop dementia with minimal loss to follow-up rates and improved completeness of diagnosis.

Demonstrating that patients with recorded dementia have an earlier onset of typical symptoms, functional impairment and death than patients in the general population would support the veracity of diagnosed dementia recorded in electronic health records and its use as an outcome or exposure in cohort studies and for evaluating policy. Previous studies have found that dementia is poorly recorded in routine clinical practice in comparison to face-to-face studies, although this varies by setting and region. However, ascertainment may be improved by examining linked, longitudinal resources. Comparing the lifetime risk of dementia calculated from linked electronic health records with lifetime risks from other sources will also be a useful information to support the use of linked electronic health records in dementia research.

Electronic health records contain information on important health transitions in patients with dementia: from the earliest stage of the illness (depression, anxiety, memory complaints); the development of cognitive impairment that manifest as loss of capacity or missed appointments; and significant functional impairment, with admission to nursing homes or hospital admission. In this study, we will assess the validity of dementia diagnoses in linked primary care, hospital and death records, by examining the timing of important health transitions in patients with recorded dementia, and estimate the lifetime risk of recorded dementia in different age and sex groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over
* Registered with a participating general practice during the study period
* Minimum one year of records prior to study entry meeting CPRD data quality criteria
* Followed on or after 1 January 1997

Exclusion Criteria:

* Patients without recorded gender
* Less than 1 year of follow-up between study entry and date of administrative censoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients registered in English general practices contributing with data to the CALIBER research platform from 1997 onward.
Sampling Method: Non-Probability Sample
Enrollment: 51000 (Estimated)
Dates: Start 2015-09; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with dementia diagnosis (any type) in primary care that also are recorded in secondary care | 10 years
Factors associated with dementia diagnosis (any type) recording in mortality data only | 10 years
  These will be estimated from multivariable logistic regression models
Symptoms associated with subsequent diagnosis of dementia | 10 years
  These will be estimated from multivariable logistic regression models
Lifetime risk of dementia (any type) | 10 years
Lifetime risk of mortality associated with dementia (any time) | 10 years
Factors associated with dementia diagnosis (any type) recording in secondary care only | 10 years
  These will be estimated from multivariable logistic regression models
Factors associated with dementia diagnosis (any type) recording in primary care only | 10 years
  These will be estimated from multivariable logistic regression models
Proportion of patients with dementia diagnosis (any type) in primary care that also are recorded in mortality data | 10 years
Proportion of patients with dementia diagnosis (any type) in secondary care that also are recorded in mortality data | 10 years

SECONDARY OUTCOMES:
Proportion of patients with Alzheimer's disease in primary care that are also diagnosed in secondary care | 10 years
Proportion of patients with vascular dementia in primary care that are also diagnosed in secondary care | 10 years
Lifetime risk of Alzheimer's disease | 10 years
Lifetime risk of vascular dementia | 10 years
Lifetime risk of mortality associated with Alzheimer's disease | 10 years
Proportion of patients with Alzheimer's disease in primary care that are also diagnosed in mortality data | 10 years
Proportion of patients with Alzheimer's disease in secondary care that are also recorded in mortality data | 10 years
Proportion of patients with vascular dementia in primary care that are also recorded in secondary care | 10 years
Proportion of patients with vascular dementia in secondary care that are also recorded in mortality data | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- London Farr Institute of Health Informatics, London, United Kingdom